CLINICAL TRIAL: NCT04568200
Title: A Prospective, Randomized Controlled Study to Evaluate the Efficacy and Safety of Durvalumab Combined With Neoadjuvant Therapy in Patients With Local Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Study of Anti-PD-L1 in Combination With Chemo(Radio)Therapy for Resectable Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69152630
Record Dates: First submitted 2020-09-15; First posted 2020-09-29 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — durvalumab; Carboplatin; Drug Therapy; Paclitaxel; Radiotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- durvalumab and neoadjuvant therapy (Experimental): durvalumab 1500mg i.v. day 1-22-43-64 Carboplatin AUC = 4-5 i.v day 1-22-43-64 Paclitaxel 75 mg/m2 i.v day 1-22-43-64 with/without Radiotherapy 23 x 1.8 Gy
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiotherapy 23 x 1.8 Gy
- normal saline and neoadjuvant therapy (Placebo Comparator): normal saline 500ml i.v. day 1-22-43-64 Carboplatin AUC = 4-5 i.v day 1-22-43-64 Paclitaxel 75 mg/m2 i.v day 1-22-43-64 with/without Radiotherapy 23 x 1.8 Gy
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiotherapy 23 x 1.8 Gy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg i.v. day 1-22-43-64
  Arms: durvalumab and neoadjuvant therapy
Drug: Carboplatin — Chemotherapy
  Other Names: Chemotherapy
Drug: Paclitaxel — Chemotherapy
  Other Names: Chemotherapy
Radiation: Radiotherapy 23 x 1.8 Gy — Radiotherapy 23 x 1.8 Gy
  Other Names: Radiotherapy

SUMMARY:
This is a study to evaluate the efficacy and safety of preoperative treatment with durvalumab combined with neoajuvant therapy (carboplatin, paclitaxel with/without radiation) in locally advanced resectable oesophageal squamous carcinoma.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the tumor response (by irRECIST) and pathological response of preoperative treatment with durvalumab combined with neoadjuvant therapy (carboplatin, paclitaxel with/without radiation).

Secondary objectives are:

To assess completion of treatment with durvalumab combined with chemotherapy with/without radiation treatment.

To assess toxicities of durvalumab in combination with chemoradiation. [Time Frame: up to 1 year] To assess completion of chemotherapy with/without radiation treatment. To assess withdrawal rate from surgery. To assess delay rate from surgery. To assess R0 resection rate. To assess post-operative complications. Progression Free Survival. [ Time Frame: up to 24 months ] Overall Survival. [ Time Frame: up to 24 months ]

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the esophagus.
* Surgical resectable (T3 or T4b, N0 or N+, M0), as determined by Endoscopic Ultra Sound (EUS),PET/CT, Esophageal MRI and enhanced CT scan of neck, thorax and abdomen.
* Tumor length longitudinal ≤ 10 cm; if larger than 10 cm, inclusion should be discussed with the principal investigator.
* 18≤Age≤75.
* Tumor does not involve gastro-esophageal junction.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematological, renal and hepatic functions defined as:

neutrophiles ≥ 1.5 x 109/L platelets ≥ 100 x 109/L alanine transaminase≤2 x upper normal limit hemoglobin ≥ 5.6 mmol total bilirubin ≤ 1.5 x upper normal limit creatinine clearance (Cockroft) ≥60 ml/min

* Written, voluntary informed consent.

Exclusion Criteria:

* Past or current history of malignancy other than entry diagnosis interfering with prognosis of esophageal cancer.
* T1, T2 tumors or in situ carcinoma.
* metastatic oesophageal cancer.
* Pregnancy (positive serum pregnancy test), planning to become pregnant, and lactation.
* Previous chemotherapy, radiotherapy, and/or treatment with checkpoint inhibitors.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) precluding major surgery.
* Pulmonary fibrosis and/or severely impaired lung function precluding major surgery.
* Pre-existing motor or sensory neurotoxicity greater than WHO grade 1.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10 mg/day prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine.
* Has an active infection requiring systemic therapy which has not resolved 3 days (simple infection such as cystitis) to 7 days (severe infection such as pyelonephritis) prior to the first dose of trial treatment.
* Has a diagnosis of acute or chronic hepatitis B, hepatitis C, known immunodeficiency or human immunodeficiency virus (HIV).
* Patients with prior allogeneic stem cell or solid organ transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
tumor response | up to 12 months
  assess the tumor response (by irRECIST) of preoperative treatment with durvalumab combined with neoadjuvant therapy
pathological response | up to 12 months
  assess the pathological response (by CAP classification) of preoperative treatment with durvalumab combined with neoadjuvant therapy

SECONDARY OUTCOMES:
Percentage completion of treatment with durvalumab combined with chemotherapy with/without radiation treatment | up to 3 months
  Percentage completion of treatment with durvalumab combined with chemotherapy with/without radiation treatment
Incidence and severity of toxicity | up to 12 months
  Incidence and severity of toxicity defined to CTCAE v4.03 and Radiation Oncology Group (RTOG) criteria
Percentage completion of chemotherapy with/without radiation treatment | up to 3 months
  Percentage completion of chemotherapy with/without radiation treatment
Percentage withdrawal rate from surgery due to durvalumab related complications | up to 3 months
  Percentage withdrawal rate from surgery due to durvalumab related complications
Percentage delay of surgery due to durvalumab related complications | up to 3 months
  Percentage delay of surgery due to durvalumab related complications
R0 resection rate | up to 3 months
  R0 resection rate
Incidence and severity of post-operative complications to the Dindo classification | up to 3 months
  Incidence and severity of post-operative complications to the Dindo classification
Progression free survival | up to 24 months
  Progression free survival
Overall survival | up to 24 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jia He, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China